CLINICAL TRIAL: NCT05777187
Title: Integration of Machine Learning and Clinical Decision Support to Prevent Postoperative Delirium in Patients with Cognitive Impairment
Brief Title: Mitigation of Postoperative Delirium in High-Risk Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment closed due to low enrollment.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of California, Los Angeles (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ira Hofer, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-22-00920; 22-00920 (Other: Advarra/CIRBI); 5U54AG063546 (NIH)
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post-operative Delirium; Decision Support Systems, Clinical; Cognitive Impairment
MeSH Terms: conditions — Emergence Delirium; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical Decision Support (Experimental): Clinical decision support alerts in the electronic health record directed towards anesthesiologists caring for patients with preexisting cognitive impairment.
  Interventions: Other: Clinical Decision Support
- Standard of Care (No Intervention): No clinical decision support will appear, and standard of care procedures will take place.

INTERVENTIONS:
Other: Clinical Decision Support — The intervention will consist of clinical decision support alerts in the electronic health record directed towards anesthesiologists caring for patients with preexisting cognitive impairment. This intervention will alert towards delirium risk informed by history of cognitive impairment and promote 12 evidence based best practices during care for perioperative patients.
  Arms: Clinical Decision Support

SUMMARY:
Among patients with cognitive impairment (CI) that undergo surgery, the risk for developing postoperative delirium (POD) is high (50%) and associated with further morbidity and mortality. Yet, 30-40% of POD cases are preventable with perioperative management. This randomized pragmatic clinical trial aims to assess incidence of POD in adult surgical patients with CI, as well as provider adherence to a set of 12 perioperative best practice recommendations for perioperative management. Electronic health record (EHR) data will be used to identify patients as high risk for developing POD and clinical decision support (CDS) prompts within the EHR will display best practices. Cases will be randomized to either the control group, usual care or the intervention which includes the high-risk alert and best practice prompts.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a history of cognitive impairment (CI) undergoing surgery at the Mount Sinai Health System.
* Attending physicians, resident physicians, and nurse anesthetists at the Mount Sinai Health System receiving CDS alerts during EHR system implementation.

Exclusion Criteria:

* Patients will be excluded if this not their first surgery since study start, if they do not have cognitive impairment based on EHR data, or if the surgery is for organ donation.
* There will be no exclusion criteria for providers or historical controls.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24426 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
4AT Delirium Score | Postoperative days 0-7
  Incidence of Postoperative Delirium measured using the 4AT delirium assessment documentation
  Scoring:
  4 or above: possible delirium +/- cognitive impairment 1-3: possible cognitive impairment 0: delirium or severe cognitive impairment unlikely (but delirium still possible if [4] information incomplete)

SECONDARY OUTCOMES:
Perioperative Best Practices proportion | Day 1
  For each of the 12 practices, adherence will be measured as a binary variable; overall protocol adherence will be defined as the proportion of the 12 practices performed by the anesthesia team.
  The 12 perioperative best practices are grouped in 5 intervention domains including, avoid potential inappropriate medication, perioperative glycemic control, avoid hypotension, maintain normothermia, and titrate anesthetic depth. Within avoid potential inappropriate medication is avoid diphenhydramine, scopolamine, and midazolam. Within perioperative glycemic control is check pre-op glucose, check glucose every 2 hours, maintain glucose <200 mg/dL, and check post-anesthesia care unit glucose. Within avoid hypotension is Mean Arterial Pressure >65 mmHg. Within maintain normothermia is use temperature probe and maintain temperature >36 degrees Celsius. Within titrate anesthetic depth is age adjusted MAC<1 and monitor anesthesia depth.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Hofer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Health System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The research team will be collecting the data in a data warehouse, but it will be extracted by an honest broker de-identified. No participant level data will be shared outside Sinai or the study team.